A Mechanistic Perspective on Post-Activation Performance
Enhancement Responsiveness: A Randomized Controlled
Study of Acute Changes in Muscle Architecture, Contractile
Property Kinetics, and Muscle Excitability
NCT06982937

15.03.2023

## Appendix No. 2

to the Regulations of the Bioethics Committee

## PARTICIPANT'S DECLARATION

| Surname and first name of the participant: |
|---|
| Age: |
| Address: |
| Name and surname of the principal investigator: Artur Terbalyan |
| Contact phone numbers for the participant: 322075368; 536899973 |
| <b>Study title:</b> Application of modern training methods to optimize selected parameters of anaerobic performance and motor abilities in team sports |
| I hereby declare that I have been informed by: Artur Terbalyan |

1. **1. I have been informed** about the aim of the intended research and the manner in which it will be conducted, and I have had the opportunity to ask the experimenter questions and have received answers to those questions. I understand what the study involves and why my consent is required. I have read the "Information for the Participant," of which I received one copy. I have been informed about the potential

| risks associated with the research prograthe medical experiment. | am. Therefore, I voluntarily consent to undergo |
|---|---|
| date and signature of the principal investigator | date and signature of the participant or legal guardian |
| 2. <b>2. I may refuse consent</b> to participate in during the procedures—and this will in r | · |
| date and signature of the principal investigator | date and signature of the participant or legal guardian |
| | ng of my data to the extent necessary to conduct prevents identification of my person by legal or in the protocol as conducting the study. |
| date and signature of the principal investigator | date and signature of the participant or legal guardian |
| about the terms of insurance covering an | participant/volunteer) I have been informed by negative consequences of participation in the en access to the insurance policy from which |
| I have received one copy of the "Participa | ant's Declaration." |
| date and signature of the principal investigator | date and signature of the participant or legal guardian |